CLINICAL TRIAL: NCT01076673
Title: Articular Cartilage Regeneration With Autologous Peripheral Blood Stem Cells Versus Hyaluronic Acid: A Randomized, Controlled Trial
Brief Title: Effect of Autologous Peripheral Blood Stem Cell Treatment on Articular Cartilage Regeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kuala Lumpur Sports Medicine Centre (Other)
Collaborators: Ministry of Science, Technology and Innovation (MOSTI) Malaysia (Unknown)
Responsible Party: Principal Investigator, Dr. Khay-Yong Saw, Consultant Orthopaedic Surgeon, Kuala Lumpur Sports Medicine Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KLSMC-001
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Articular Cartilage Disorder of Knee
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PBSC and Hyaluronic Acid (Experimental): Peripheral blood stem cells and hyaluronic acid injections
  Interventions: Biological: Peripheral blood stem cells and hyaluronic acid injections
- Hyaluronic Acid (Active Comparator): Hyaluronic Acid
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Biological: Peripheral blood stem cells and hyaluronic acid injections — Peripheral blood stem cells and hyaluronic acid injections
  Other Names: PBSC and HA
  Arms: PBSC and Hyaluronic Acid
Drug: Hyaluronic Acid — Hyaluronic acid injections
  Other Names: HA
  Arms: Hyaluronic Acid

SUMMARY:
The purpose of this study was to compare histologic and MRI evaluation of articular cartilage regeneration in patients with chondral lesions treated by arthroscopic subchondral drilling followed by postoperative intra-articular injections of hyaluronic acid (HA) with and without peripheral blood stem cells (PBSC)

DETAILED DESCRIPTION:
The purpose of this study was to compare histologic and magnetic resonance imaging (MRI) evaluation of articular cartilage regeneration in patients with chondral lesions treated by arthroscopic subchondral drilling followed by postoperative intra-articular injections of hyaluronic acid (HA) with and without peripheral blood stem cells (PBSC)

ELIGIBILITY:
Inclusion Criteria:

* Patients who have signed informed consent form
* Patients with only unilateral isolated or multiple knee articular cartilage lesions demonstrated MRI scanning, with up to one previous operation on that knee
* Patients who are either male or female aged between 18 to 50 years old, corresponding to availability of normative International Knee Documentation Committee (IKDC) data.
* Female patients of childbearing age must have negative pregnancy tests and are advised to take contraceptive precautions throughout the study.

Exclusion Criteria:

* Patients with bilateral knee lesions
* Patients with the presence of ligamentous injury which would require reconstruction, varus or valgus deformity greater than 10 degrees, previous open total menisectomy requiring osteotomy, and cases that require complex surgery prior to cartilage regeneration
* Patients with significant cognitive impairment, non-ambulatory status or lower extremities amputation other than toes, serious illness or medication affecting operative risk or wound healing (e.g. steroid intake, anticoagulation), and poorly controlled diabetes mellitus with a baseline HbA1c more than 8
* Patients with significant peripheral vascular disease as indicated by absent dorsalis pedis or posterior tibial pulses.
* Patients who cannot read English will be excluded from the study as they will be unable to complete the study questionnaires in an objective manner
* Female patients who are pregnant
* Patients with any contradictions to MRI scanning
* Patients with body mass index (BMI) of over 35

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in tissue histology after subchondral drilling surgery using serial MRI scanning and cartilage biopsies | 18 months

SECONDARY OUTCOMES:
Improved long term functional outcome of subchondral drilling surgery in the knee joint | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Khay-Yong Saw, Dr., Principal Investigator — Kuala Lumpur Sports Medicine Centre
Locations (1):
- Kuala Lumpur Sports Medicine Centre, Kuala Lumpur, Malaysia

REFERENCES:
- [Result] Saw KY, Anz A, Siew-Yoke Jee C, Merican S, Ching-Soong Ng R, Roohi SA, Ragavanaidu K. Articular cartilage regeneration with autologous peripheral blood stem cells versus hyaluronic acid: a randomized controlled trial. Arthroscopy. 2013 Apr;29(4):684-94. doi: 10.1016/j.arthro.2012.12.008. Epub 2013 Feb 4. PMID 23380230